CLINICAL TRIAL: NCT02931695
Title: Influence of Sex Hormones Variation During Third Trimester of Pregnancy and Post-partum on QT Interval Duration
Acronym: QuTe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: INSERM 1166 ICAN UPMC (Unknown); CIC1901-Centre d'Investigation Clinique Paris-Est (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 2016-01
Record Dates: First submitted 2016-09-15; First posted 2016-10-13 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy
Keywords: post partum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregnant women (Other): Women during third trimester of pregnancy and in the first trimester of post partum
  * ECG
  * circulating sex hormones levels
  Interventions: Other: evaluation of QT interval duration; Other: circulating sex hormones levels sample
- women in the first trimester of post partum (Other): Women (same in first arm) in the first trimester of post partum
  * ECG
  * circulating sex hormones levels
  Interventions: Other: evaluation of QT interval duration; Other: circulating sex hormones levels sample

INTERVENTIONS:
Other: evaluation of QT interval duration — ECG to evaluation of QT interval duration
Other: circulating sex hormones levels sample — Association between circulating sex hormones levels (progesterone, estradiol, testosterone, FSH) and QTcF duration (univariate and multivariate analysis).

SUMMARY:
QT interval prolongation, corrected for heart rate (QTc), either spontaneous or drug-induced, is associated with an increased risk of torsades de pointes and sudden death. Women are at higher risk of torsades de pointes, particularly during post-partum and the follicular phase.

The aim of this study is to explore if QTc duration is prolonged during post-partum as compared to the 3rd trimester of pregnancy

DETAILED DESCRIPTION:
Sex steroid hormones are known to influence heart repolarization. Overall, estradiol is considered to promote QTc lengthening while progesterone and testosterone shorten QTc. New findings suggest more complex regulation of QTc by sex steroid hormones involving also follicle-stimulating hormone, which is associated to prolongation of QTc. Another important aim of this study is to study the influence of sex hormones on QTc duration.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 yo) pregnant women in their third trimester
* Able to give her consent

Exclusion Criteria:

* Concomitant intake of QTcF prolonging drugs
* Past medical history of cardiovascular or endocrino-metabolic conditions (except hypertension or diabetes)
* QRS >120 msec on electrocardiogram

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Difference in QTcF duration (Corrected for heart rate according to Fridericia method) between third trimester of pregnancy and post-partum. | third trimester of pregnancy and 3 to 6 months delivery

SECONDARY OUTCOMES:
Association between circulating sex hormones levels (progesterone, estradiol, testosterone, FSH) and QTcF duration (univariate and multivariate analysis). | third trimester of pregnancy and 3 to 6 months delivery

CONTACTS AND LOCATIONS:
Overall Officials: Joe-Elie SALEM, MD PHD, Principal Investigator — Centre d'investigation Clinique - Paris est
Locations (1):
- Centre d'investigation Clinique - Paris est, Paris, France